CLINICAL TRIAL: NCT04859673
Title: Influence of Radial Extracorpeal Shock Wave Therapy on Sonographic Findings in Patients With Hemiplegic Shoulder Pain
Brief Title: Influence of Radial Extracorpeal Shock Wave in Hemiplegic Shoulder Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Ibrahim Ahmed Ibrahim Abu Ella, assistant lecturer, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002870
Record Dates: First submitted 2021-04-13; First posted 2021-04-26 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Hemiplegia; Spastic
Keywords: Sonography; Pain
MeSH Terms: conditions — Hemiplegia; Muscle Spasticity; Pain

STUDY DESIGN:
Intervention Model Description: The selected patients will be randomly assigned to two equal groups (study group (GI), and control group (GII).The study group (GI) will be treated by the radial extracorporeal shock wave in addition to design physical therapy program.
  • The control group (GII) will be treated by sham radial extracorporeal shock wave in addition to the same design physical therapy program of (GI).
Who Masked: Participant
Masking Description: The patients in control group will be treated by sham radial extracorporeal shock wave therapy in addition to, the same design physical therapy program. Stimulation will not deliver as the transmitter head will be removed.
  The patients will receive the same frequency of air pressure and sound
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): Patients will received 3,000 pulses, 1,500 pulses per site at a frequency of 12 Hz per session with the submaximal pressure between 0.39 and 1.95 mJ/mm2 (1.0 and 5.0 bar), depending on the level which the patient can tolerate without local anesthetics.
  Interventions: Device: radial extracorpeal shock wave
- control group (Sham Comparator): The patients in this group will be treated by sham radial extracorporeal shock wave therapy. Stimulation will not deliver as the transmitter head will be removed. The patients will receive the same frequency of air pressure and sound
  Interventions: Device: radial extracorpeal shock wave

INTERVENTIONS:
Device: radial extracorpeal shock wave — Swiss DolorClast® Master - Shockwave Therapy System will be used to apply the radial extracorporeal shock wave. It consists of master console, Evo Blue hand-piece, 15mm and 36mm interchangeable contact heads (applicators), contact gel, cart, and external compressor

SUMMARY:
The purposes of this study are to examine sonographic structural changes pre and post the radial extracorporeal shock wave intervention in hemiplegic shoulder pain, and to assess the relationships between sonographic structural changes and hemiplegic shoulder pain.

DETAILED DESCRIPTION:
Painful shoulder is a common complication following hemiplegic stroke. This pain may interfere with functional improvement, the patient's quality of life, and it may impede the process of rehabilitation. Further understanding of rotator cuff tendon impairment and other shoulder soft tissue structural abnormalities in stroke patients may help clinicians in assigning more complete therapeutic plans to hemiplegic patients. The radial extracorporeal shock wave therapy has promising results in patients with musculoskeletal problems and in those with various causes of HSP, including spasticity, rotator cuff problems, adhesive capsulitis, and complex regional pain syndrome .The purposes of this study are to examine sonographic structural changes pre and post the radial extracorporeal shock wave intervention in hemiplegic shoulder pain, as well as to explore the relationships between sonographic structural changes and hemiplegic shoulder pain. This study will be a benefit in the physical therapy field and may guide rehabilitation programs of physical therapy towards better results through decreasing time needed to perform activity of daily living, decreasing dependency and making patient an active member in society.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient's age ranges from 40 to 60 years. 2. Spasticity of upper limb ranges from mild to moderate (grade 1+: 2) according to modified aschworth scale (MAS).

  3. Patients with sufficient cognitive abilities that enables them to understand and follow instructions (Mini-Mental Scale >24).

  4. Patient who understand the study process and signed the informed consent form.

  5. Patient with stroke more than 3 months ago. 8. Patient with shoulder pain and limited range of motion (ROM) or loss of motion in the proximal arm on the hemiplegic side.

Exclusion Criteria:

* The following patients will be excluded from the study:

  1. Patients who cannot express their own pain intensity.
  2. Patients with a history of trauma or surgery to the shoulder on the affected side.
  3. Patients with history of oral NSAIDs 3 days before this study or take warfarin medication with an international normalized ratio above 4.0.
  4. Patients with a history of shoulder pain before the stroke.

  6. Patients who have received a previous shoulder intra-articular injection or other interventions on the affected shoulder within one month before rESWT.

  7. Patients with cardiac pacemaker. 8. Patients who have osteoporosis. 9. Patients with psychological problems.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of hemiplegic shoulder structural changes by ultrasonography | Baseline
  Ultrasonography evaluation includes long head of biceps tendon ,subscapularis tendon, supraspinatus tendon, infraspinatus tendon. Each abnormal ultrasound (US) finding will be assigned a score of one (1) if present or zero (0) if absent. Long head of biceps effusion, sub acromial sub deltoid bursa effusion, subluxation, and adhesive capsulitis scored. Tendon tear, tendinosis, and tendon degeneration will be similarly scored for each of the four examined tendons per shoulder. The sum of these scores yielded a raw ultrasound (US) score; such that the minimum score was zero (normal examination) while the maximum score amounted to sixteen .The raw US scores will be further grouped into graded US scores, such that scores of 0, 1-2, 3-4, 5-6, and more than 6 abnormal sonographic findings represented normal shoulder, mild damage, moderate damage, severe damage, and intense damage, respectively

SECONDARY OUTCOMES:
Pain assessment by using shoulder pain and disability index (SPADI). | Baseline
  Shoulder pain and disability index is a shoulder specific self-reported questionnaire measuring pain and disability in patients with shoulder pain. It contains 5 items assessing pain and 8 items assessing shoulder function. Each item is scored on visual analogue scale with (Right end) defined as "worst pain imaginable/ so difficult required help", (Left end)"no pain/no difficulty". Scores will be calculated as follow, in part one pain scores in all questions will be added, and the mean value will be chosen. In part two functional scores of all questions will add and the mean value will be chosen for the purpose of data analysis. Final score for each part will be statistically analyzed separately

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim A Abu-Ella, MSC, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wilson RD, Chae J. Hemiplegic Shoulder Pain. Phys Med Rehabil Clin N Am. 2015 Nov;26(4):641-55. doi: 10.1016/j.pmr.2015.06.007. Epub 2015 Sep 9. PMID 26522903